CLINICAL TRIAL: NCT05508347
Title: Sichuan Cancer Hospital and Institute, Sichuan Cancer Center, School of Medicine, University of Electronic Science and Technology of China
Brief Title: Nituzumab (Taixinsheng ®） A Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Study on the Efficacy and Safety of Combined Induction Chemotherapy for Locally Advanced Nasopharyngeal Carcinomatreatment of Locally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Mei Feng, Chief physician, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ahead-NC-202203
Record Dates: First submitted 2022-08-14; First posted 2022-08-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): 3 cycles of docetaxel combined with cisplatin induction chemotherapy combined with 9 times of 200mg nituzumab targeted therapy, and sequential 2-3 cycles of concurrent chemoradiotherapy based on cisplatin chemotherapy combined with 7 times of nituzumab targeted therapy.
  Interventions: Drug: Nituzumab/placebo
- control group (Placebo Comparator): 3 cycles of docetaxel combined with cisplatin induction chemotherapy combined with 9 times of placebo treatment, and sequential 2-3 cycles of concurrent chemoradiotherapy based on cisplatin chemotherapy combined with 7 times of nituzumab targeted therapy
  Interventions: Drug: Nituzumab/placebo

INTERVENTIONS:
Drug: Nituzumab/placebo — Test group: 3 cycles of induction chemotherapy combined with 9 times of nituzumab targeted therapy followed by 2-3 cycles of synchronous radiotherapy and chemotherapy combined with 7 times of nituzumab targeted therapy, a total of 16 times of nituzumab targeted therapy, equivalent to the whole course targeted therapy.
  Control group: 3 cycles of induction chemotherapy combined with 9 times of placebo treatment followed by 2-3 cycles of concurrent chemoradiotherapy combined with 7 times of nituzumab targeted therapy, a total of 7 times of nituzumab targeted therapy, only targeted therapy during concurrent chemoradiotherapy
  Other Names: Nituzumab injection (taixinsheng)

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a head and neck tumor. Studies have shown that more than 70% of patients are diagnosed with locally advanced nasopharyngeal carcinoma at the time of initial diagnosis. The 3-year survival rate of locally advanced nasopharyngeal carcinoma after chemotherapy is over 90%, but 30% of patients still have recurrence and distant metastasis. Therefore, while improving the level of radiation therapy technology, we should study multidisciplinary comprehensive treatment methods and put forward the biological concept of "cure". Induction chemotherapy can effectively create better radiotherapy conditions for locally advanced nasopharyngeal carcinoma, especially for patients with large lesions, improve the treatment response rate, and may reduce the local recurrence and distant metastasis rate. After the end of neoadjuvant chemotherapy, compared with patients who only reached SD, patients who reached CR had a significant survival benefit; Other patients had a reduced rate of distant metastasis, which aroused our interest, although there was no obvious survival benefit. The national multicenter phase II clinical study showed that nitumab combined with radiotherapy significantly improved the 3-year survival rate of patients with locally advanced nasopharyngeal carcinoma compared with radiotherapy alone. According to the previous related research results, nitumab combined with induction chemotherapy or concurrent chemoradiotherapy has a certain effect on nasopharyngeal carcinoma without obvious adverse reactions. However, prospective studies on the short-term efficacy and safety of local advanced nasopharyngeal carcinoma combined with induction chemotherapy and concurrent chemoradiotherapy are still lacking (Taisheng ®）。

DETAILED DESCRIPTION:
In recent years, studies have found that epidermal growth factor (EGF) is related to the proliferation of tumor cells, and a lot of evidence shows that the overexpression of epidermal growth factor receptor (EGFR) is related to the formation of metastases and poor prognosis. The expression rate of EGFR in nasopharyngeal carcinoma is 68%-89%. Therefore, the EGF/EGFR system may become a new therapeutic target for the treatment of head and neck squamous cell carcinoma, and the monoclonal antibody binding to the receptor becomes a potentially effective anticancer biological agent. The effect of radiotherapy to achieve the effect of inhibiting the growth of cancer cells. It is much higher than other solid tumors and is closely related to the prognosis of patients with nasopharyngeal carcinoma. A retrospective paired analysis by Peng et al suggested that induction chemotherapy combined with anti-EGFR receptor therapy may be a more effective strategy for locally advanced nasopharyngeal carcinoma following IMRT. Nimotuzumab (Taixinsheng®) is a recombinant humanized monoclonal antibody against EGFR jointly developed by Baitai Biopharmaceutical Co., Ltd. and Cuban Center for Molecular Immunology, and has been listed in 19 foreign countries. Nimotuzumab is a humanized monoclonal antibody that can competitively inhibit the binding of endogenous ligands to EGFR, block the downstream signal transduction pathway mediated by EGFR, thereby inhibiting tumor cell proliferation and promoting tumor cell apoptosis , inhibit angiogenesis and increase the sensitivity of radiotherapy and chemotherapy; due to the characteristics of humanization and high selectivity, compared with cetuximab, nimotuzumab has fewer adverse reactions and a lower incidence of rash. At present, phase I and II clinical studies of Nimotuzumab (Taixinsheng®) combined with radiotherapy in the treatment of advanced nasopharyngeal carcinoma have been completed in China, and have been approved by the SFDA. A national multicenter phase II clinical study showed that compared with radiotherapy alone, nimotuzumab combined with radiotherapy significantly improved the 3-year OS of patients with locally advanced nasopharyngeal carcinoma (77.61% vs. 84.3%, P<0.05). Therefore, in April 2009, Nimotuzumab entered the Chinese version of the NCCN Head and Neck Cancer Guidelines.

Regarding the efficacy of nimotuzumab during concurrent chemoradiotherapy, Shi Xingyuan et al. conducted a prospective clinical trial in 2016. The control group was treated with concurrent chemoradiotherapy (chemotherapy single-agent cisplatin), and the experimental group was treated with concurrent chemoradiotherapy based on the treatment of the control group. Combined with nimotuzumab, the short-term and long-term efficacy and toxic and adverse reactions of nimotuzumab combined with cisplatin concurrent chemotherapy in the treatment of locally advanced (III-IVB stage) nasopharyngeal carcinoma were observed. The results showed that in the experimental group compared with the control group, the ORR was 100% VS.91.67% (p<0.05) at 3 months after treatment, the CR rate at 3 months after treatment was 91.7% VS.79.3% (p<0.05), and the 5-year OS was 87.5 % VS.62.5%, (P=0.036), the incidence of adverse reactions was basically the same (P>0.05). In 2018, Wang retrospectively analyzed 1104 patients with stage III-IVB nasopharyngeal carcinoma, all of whom received concurrent chemoradiotherapy after induction chemotherapy, with or without nimotuzumab. Induction chemotherapy followed by concurrent chemoradiotherapy and nimotuzumab was effective and well tolerated in the treatment of locally advanced nasopharyngeal carcinoma, with a 5-year OS of 94.5% vs. 85.6% in the control group (P= 0.058), PFS 87.4 % vs. 81.3% (P=0.225), and the 5-year DMFS was 95.8% vs. 83.9% (P=0.007), respectively, indicating that concurrent chemoradiotherapy and nimotuzumab could achieve the best survival benefit after induction chemotherapy.

In the past, studies on the application of nimotuzumab during induction chemotherapy were carried out. In 2014, Song et al. conducted a prospective clinical study. A total of 168 patients with nasopharyngeal carcinoma (stage II-IV) received 2-3 cycles of induction chemotherapy (IC). ) followed by concurrent chemoradiotherapy (CCRT), of which 56 patients were added with Nimotuzumab (Nimo) and were divided into three groups: A, IC + CCRT; group B: IC (with Nimotuzumab) + CCRT; group C: IC + CCRT (Nimotuzumab added at the same time). IC+Nimo,+CCRT VS. IC+CCRT 5-year OS were 93.0% VS. 74.8%, P=0.038, IC+Nimo,+CCRT VS. IC+CCRT 5-year PFS rates were 89.3% VS. .72.7% (P=0.144). There were no significant adverse reactions in the nimotuzumab treatment group. The 5-year OS and PFS of group C were 80.4 ± 7.9% and 76.4 ± 8.5%, respectively, which were not statistically significant compared with group A (p = 0.257 and p = 0.611, respectively). In 2019, Lu Ying et al. conducted a multi-center clinical study, including 58 patients in the III-IVB NPF group (Nimotuzumab combined with PF regimen induction therapy group) and 60 TPF patients (docetaxel, cisplatin, fluorouracil regimen induction therapy group) Chemotherapy group), after 2 cycles of induction therapy, all patients received cisplatin concurrently with intensity-modulated radiation therapy (IMRT). The safety and short-term efficacy of the two groups were compared. In the induction stage, the ORR NPF VS.TPF of cervical lymph nodes and nasopharyngeal primary lesions were 70.69% VS. 0.05). Compared with the TPF group, induction therapy in the NPF group had a more significant effect on cervical lymph nodes (81% vs. 60% P=0.036). There was no significant difference in efficacy evaluation (P>0.05). During induction therapy, neutropenia and gastrointestinal reactions were significantly improved compared with TPF group (P=0.028, P=0.049). During the concurrent chemoradiotherapy phase, compared with the TPF group, the gastrointestinal reaction, oral mucositis and radiodermatitis in the NPF group were significantly improved (P=0.038, P=0.041, P=0.035). It shows that for locally advanced nasopharyngeal carcinoma receiving cisplatin concurrent IMRT, induction therapy with nimotuzumab combined with PF regimen has better lymph node remission rate and milder adverse reactions; the patient is resistant to subsequent concurrent chemoradiotherapy The receptivity is better, but the long-term efficacy needs further follow-up observation.

In addition, Zhao Chong et al. conducted an open-label, multi-center, phase II clinical trial to explore the efficacy and adverse reactions of cisplatin and 5-fluorouracil combined with nimotuzumab in the treatment of metastatic nasopharyngeal carcinoma after previous treatment. In this study, PF chemotherapy The objective response rate of patients in the combined nimotuzumab treatment group was 71.4%, the disease control rate was 85.7%, and the median progression-free survival time was 6.47 months, which was longer than that of the PF chemotherapy group alone in the phase III study during the same period (patients in the PF chemotherapy group). The objective response rate was 42%, and the median progression-free survival was 5.6 months), and in patients who received ≥12 doses of nimotuzumab-targeted therapy, the objective response rate was 92.6%, and the median progression-free survival was 92.6%. The time was 7.29 months, and the curative effect was significantly better than that of PF chemotherapy alone or GP chemotherapy group.

Based on the results of previous relevant studies, nimotuzumab combined with induction chemotherapy or concurrent chemoradiotherapy has a certain curative effect on nasopharyngeal carcinoma, and there are no significant adverse reactions. However, there is currently a lack of prospective application research data on the short-term efficacy and safety of nimotuzumab (Taixinsheng®) combined with induction chemotherapy and concurrent chemoradiotherapy in the treatment of locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion criteria:

1. Voluntarily participate and sign the informed consent in writing.
2. Age: 18-70 years old, gender is not limited.
3. Nasopharynx squamous cell carcinoma diagnosed by histopathology.
4. Nasopharyngeal carcinoma 2018 AJCC (Eighth Edition) staging: t2-4n2m0 (metastatic lymph nodes have one of the following risk factors: the shortest length of the largest lymph node is ≥ 3cm or the lymph node is liquefied and necrotic or the lymph node envelope is invaded) or t1-4n3m0.
5. Immunohistochemistry: EGFR (+).
6. The primary tumor can be measured.
7. Kaplan score > 70.
8. Survival expectation ≥ 6 months.
9. Women in childbearing period should ensure to take effective contraception during the study period.
10. Hemoglobin (Hgb) ≥ 90 g / L, white blood cell (WBC) ≥ 4 × 109 / L, platelet (PLT) ≥ 90 × 109 /L.
11. Liver function: ALT and / or ast < 1.5 times the upper limit of normal value (ULN), and TBIL < 1.5 times the upper limit of normal value (ULN).

Renal function: serum creatinine < 1.5 times the upper limit of normal value (ULN); Creatinine clearance rate shall not be lower than 60ml / min.

Exclusion criteria：

1. There is evidence of distant metastasis.
2. The primary tumor or lymph node has been treated surgically (except biopsy).
3. Patients with primary focus or lymph nodes who have received radiotherapy.
4. Those who have received epidermal growth factor targeted therapy.
5. The primary lesion has received chemotherapy or immunotherapy.
6. Have had other malignant tumors (except non melanoma skin cancer or cervical carcinoma in situ).
7. Subjects who have received other drug tests in the past 1 month.
8. > grade I peripheral neuropathy.
9. Pregnant or lactating women and women of childbearing age who refuse contraception during the treatment observation period.
10. Those with severe allergic history or special constitution.
11. A history of severe lung or heart disease.
12. Known to be infected with HIV virus or active viral hepatitis.
13. Received live vaccine within 30 days of the planned start of study drug treatment.
14. Those who refuse or cannot sign the informed consent form.
15. Drug or alcohol addicts.
16. Persons with personality or mental illness, without or with limited capacity for civil conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate after induction treatment period | 2 months after the start of treatment
  Complete remission (CR) rate within 5 days before the start of concurrent chemoradiotherapy after 3 cycles of induction chemotherapy

SECONDARY OUTCOMES:
Objective response (ORR) rate | 3 months after the start of treatment
  Objective response (ORR) rate within 5 days before the start of concurrent chemoradiotherapy after induction chemotherapy;
The tumor regression rate (TRR) | 2 months after the start of treatment
  The tumor regression rate (TRR) after induction therapy was evaluated within 5 days before the start of concurrent chemoradiotherapy;
Objective remission (ORR) | 2 months after the start of treatment
  Objective remission (ORR) rate within 5 days and at the third month after the end of concurrent chemoradiotherapy;
Complete remission (CR) rate | 3 months after the start of treatme
  Complete remission (CR) rate within 5 days and at the third month after the end of concurrent chemoradiotherapy;
disease-free survival (DFS) rate | 3, 5-year
  3, 5-year disease-free survival (DFS) rate
overall survival (OS) rate | 3, 5-year
  3, 5-year overall survival (OS) rate
regional recurrence free survival (lrrfs) rate | 3, 5-year
  3, 5-year regional recurrence free survival (lrrfs) rate
distant metastasis free survival (DMFS) rate | 3, 5-year
  3, 5-year distant metastasis free survival (DMFS) rate

CONTACTS AND LOCATIONS:
Overall Officials: MEI FENG, doctor, Principal Investigator — 四川省肿瘤研究所
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No